CLINICAL TRIAL: NCT05233969
Title: An Investigation of Factors Affecting Pain-Related Self-Efficacy in Individuals With Chronic Neck Pain
Brief Title: Pain-Related Self-Efficacy in Individuals With Chronic Neck Pain
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, MERVE KARAPINAR, Research Assistant, Physiotherapist, Hacettepe University
Other Study IDs: 326
Record Dates: First submitted 2022-02-01; First posted 2022-02-10 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Neck Pain
Keywords: Neck Pain; Self Efficacy; Physical Activity
MeSH Terms: conditions — Neck Pain; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The factors affecting pain-related self-efficacy in individuals with chronic neck pain were investigated. A total of 69 subjects participated in the study. After the demographic data of the subjects were taken, pain-self-efficacy questionnaire, Timed Up and Go Test, Berg Balance Scale and International Physical Activity Questionnaire were administered, respectively.

ELIGIBILITY:
Inclusion Criteria;

1. Adults aged 30 to 65 years,
2. Adults with neck pain for at least 3 months,
3. Having a score of 3 or more on the visual analog scale for pain ,
4. To be willing to participate in the study.

Exclusion Criteria;

1. Diagnosed with neurological, vestibular, rheumatic, or endocrine disorders,
2. Had previous spinal surgery, neck trauma associated with post-traumatic amnesia or concurrent head injury, or cervical fracture or dislocation,
3. currently receiving treatment for neck pathology.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with chronic neck pain
Sampling Method: Probability Sample
Enrollment: 69 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-03-20 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Pain-Self-Efficacy Questionnaire(PSEQ) | five minutes
  The Pain Self-Efficacy Questionnaire is composed of 10 items assessing the patient's self-efficacy beliefs on performing a range of life activities taking pain into consideration. Each item is rated on a 7-point Likert scale ranging from 0 = not at all confident to 6 = completely confident. The maximum possible score is 60. A high Pain Self-Efficacy Questionnaire score indicates a high level of belief in one's self-efficacy in performing life activities despite experiencing pain.

SECONDARY OUTCOMES:
Time Up and Go(TUG) | five minutes
  Patients were required to stand up from a chair with armrests, walk 3 meters, turn around, return to the chair and sit down as fast as possible. The time taken to complete this task was recorded in seconds with a stopwatch. Three trials were recorded per patient and the mean time to perform the task was calculated for each patient. The mean time interval between each trial was 1 minute.
Berg Balance Scale(BBS) | ten minutes
  The BBS26 is a functional balance measurement and consists of 14 items. Each item is a 5-point ordinal scale ranging from 0 to 4, with 0 indicating an inability to complete the task entirely and 4 indicating an ability to complete the task criterion. Scores can range from 0 to 56. The higher the score, the better the balance.
International Physical Activity Questionnaire(IPAQ) | ten minutes
  The IPAQ is used to assess habitual physical activitiy during the past 7 days. The IPAQ used in the present study is the long version which covers four domains of physical activity: occupational (7 items), transportation (6 items), household/gardening (6 items) and leisure-time activities (6 items). The questionnaire also includes two questions about the time spent on sitting as an indicator of sedentary behavior. The number of days per week and the time spent on walking per day as well as moderate and vigorous activities from all four domains are recorded. The IPAQ data were converted to metabolic equivalent scores (MET-min-week-1) for each type of activity, by multiplying the number of minutes dedicated to each activity class by the specific MET score for that activity. Physical activity levels were also classified into three categories: inactive, minimally active and health-enhancing physically active, according to the scoring system provided by the IPAQ.

CONTACTS AND LOCATIONS:
Locations (1):
- Merve Karapinar, Isparta, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No